CLINICAL TRIAL: NCT00830193
Title: N-Acetylcysteine in Critically Ill Patients Undergoing Contrast Enhanced Computed Tomography: A Randomized Trial
Brief Title: N-Acetylcysteine in Critically Ill Patients Undergoing Contrast Enhanced Computed Tomography
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Martin, Claudio M., M.D. (Individual); Fran Priestap (Unknown)
Responsible Party: Dr. Claudio Martin, London Health Sciences Centre - Victoria Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LHRI-000001
Record Dates: First submitted 2009-01-13; First posted 2009-01-27 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Contrast Induced Nephropathy; Critically Ill
Keywords: N-acetylcysteine; prevention; contrast-induced nephropathy; critically ill adults
MeSH Terms: conditions — Critical Illness | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-acetylcysteine (Active Comparator): Intravenous fluid administration was administered as soon as possible following randomization (not to exceed 12 hours prior to anticipated contrast exposure) and continued for 12 hours post CT. Patients randomized to the experimental arm received intravenous normal saline plus NAC 10 grams IV (5 g pre and 2.5 g at 6 and 12 hours post-exposure) for a total of 3 doses.
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Intravenous fluid administration was administered as soon as possible following randomization (not to exceed 12 hours prior to anticipated contrast exposure) and continued for 12 hours post CT. Medication packages were prepared and dispensed by pharmacy and included three premixed and prepackaged minibags containing either 5 g in 100 cc D5W (pre-CT dose) or 2.5 g in 50 cc D5W (post-CT doses). The placebo was D5W and was colour and consistency matched by pharmacy. Patients randomized to placebo received intravenous normal saline plus 3 doses of placebo.
  Interventions: Drug: D5W Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — Medication packages were prepared and dispensed by pharmacy and included three premixed and prepackaged minibags containing either 5 g of NAC or placebo in 100 cc D5W (pre-CT dose) or 2.5 g of NAC or placebo in 50 cc D5W (post-CT doses).
  Other Names: Mucomyst
  Arms: N-acetylcysteine
Drug: D5W Placebo — Medication packages were prepared and dispensed by pharmacy and included three premixed and prepackaged minibags containing either 5 g of NAC or placebo (D5W) in 100 cc D5W (pre-CT dose) or 2.5 g NAC or placebo in 50 cc D5W (post-CT doses).
  Other Names: D5W
  Arms: Placebo

SUMMARY:
Critically ill patients frequently undergo contrast enhanced computed tomography (CT) to establish diagnoses and direct management. Contrast agents can disturb kidney function and result in kidney dysfunction. The investigators investigated the effects of high dose N-acetylcysteine (NAC) or placebo, in addition to hydration, in preventing kidney dysfunction following contrast enhanced CT) in critically ill adults in the intensive care units of two teaching hospitals.

DETAILED DESCRIPTION:
Potential participants were identified by staff intensivists or resident physicians following admission to participating ICUs. We included critically ill adult patients at least 18 years of age who consented to participate in the trial, had central venous access and a foley catheter, required a contrast-enhanced CT of any organ system(s), and were considered 'at risk' for the development of CIN. We defined 'at risk' to include patients with at least one of the following at the time of randomization (i) a serum creatinine of > 106 µmol/L and or urea > 6 mmol/L, (ii) urine output of < 0.5 cc/kg over > 4 hrs or (iii) an increase in serum creatinine of > 50 µmol/L in < 24 hours. We stratified based on the presence or absence of diabetes defined as a history of treatment with oral hypoglycemics or insulin.

We excluded patients with a (i) CK > 5,000 or the presence of myoglobinuria, (ii) a known allergy or hypersensitivity reaction to radiographic contrast dye or NAC, (iii) serious illness with imminent threat of dying (low likelihood of survival within 48-hours) or poor prognosis, (iv) pregnancy, (v) patients with cardiogenic shock (NYHA class 3 or 4 symptoms), (vi) known or suspected nephritic, nephrotic or pulmonary-renal syndromes, (vii) a post renal etiology of renal impairment, (viii) previous renal transplant, (ix) known solitary kidney, (x) serum creatinine > 200 µmol/L or (xi) recent exposure to radiographic contrast within 14 days of randomization.

The primary outcome for the study was the development of CIN defined as a rise in serum creatinine of > 50 µmol/L from the time of randomization up to day 5 following contrast exposure.

Secondary outcomes included ICU and hospital length of stay, ICU and hospital mortality and the requirement for renal replacement therapy. We recorded compliance with assigned treatment and assessed for development of severe unexpected adverse events defined as hypotension, bronchospasm and anaphylactic reactions.

ELIGIBILITY:
Inclusion Criteria:

* The investigators included critically ill adult patients at least 18 years of age who consented to participate in the trial, had central venous access and a foley catheter, required a contrast-enhanced CT of any organ system(s), and were considered 'at risk' for the development of CIN.
* The investigators defined 'at risk' to include patients with at least one of the following at the time of randomization (i) a serum creatinine of > 106 µmol/L and or urea > 6 mmol/L, (ii) urine output of < 0.5 cc/kg over > 4 hrs or (iii) an increase in serum creatinine of > 50 µmol/L in < 24 hours.

Exclusion Criteria:

* The investigators excluded patients with a

  * CK > 5,000 or the presence of myoglobinuria
  * a known allergy or hypersensitivity reaction to radiographic contrast dye or NAC
  * serious illness with imminent threat of dying (low likelihood of survival within 48-hours) or poor prognosis
  * pregnancy
  * patients with cardiogenic shock (NYHA class 3 or 4 symptoms)
  * known or suspected nephritic, nephrotic or pulmonary-renal syndromes
  * a post renal etiology of renal impairment
  * previous renal transplant
  * known solitary kidney
  * serum creatinine > 200 µmol/L or (xi) recent exposure to radiographic contrast within 14 days of randomization.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2002-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome for the study was the development of CIN defined as a rise in serum creatinine of > 50 µmol/L from the time of randomization up to day 5 following contrast exposure. | 5 days

SECONDARY OUTCOMES:
ICU length of stay | ICU stay
Hospital length of stay | Hospital stay
ICU mortality | ICU stay
Hospital Mortality | Hospital stay
Requirement for Renal Replacement Therapy | ICU

CONTACTS AND LOCATIONS:
Overall Officials: Claudio M Martin, MD, FRCPC, MSc, Study Director — London Health Sciences Centre - Victoria Hospital
Locations (2):
- Canada (2):
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - London Health Sciences Centre - University Hospital Campus, London, Ontario